CLINICAL TRIAL: NCT03177538
Title: Open Randomized Study Comparing Clinical Efficacy of Corifollitropin Alfa (Elonva) in Combination With Menotropin (Merional) With Follitropin and Lutropin Alfa (Pergoveris) for Ovarian Stimulation in Expected Suboptimal Responders
Brief Title: Corifollitropin Alfa Combined With Menotropin Versus Follitropin and Lutropin Alfa in Expected Suboptimal Responders
Acronym: TEMPER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology (Other)
Responsible Party: Principal Investigator, Valeria Muller, PhD, MD, D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001 (TEMPER-1)
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Infertility, Female
Keywords: suboptimal response; Corifollitropin alfa; IVF; Ovarian stimulation
MeSH Terms: conditions — Infertility, Female | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Menotropins; hMG-IBSA; follitropin alfa; Luteinizing Hormone, beta Subunit; pergoveris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corifollitropin alfa and menotropin (Active Comparator): Elonva 150 mcg, Merional 150-300 IU
  Interventions: Drug: Corifollitropin alfa and menotropin
- Follitropin alfa and lutropin alfa (Active Comparator): Pergoveris 300 IU
  Interventions: Drug: Follitropin alfa and lutropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa and menotropin — Procedure: Ovarian stimulation is performed by the combination of a single Corifollitropin alfa 150 mcg injection on menstrual cycle day 2-3 and daily menotropin administration at the dose of 150 IU from stimulation day 1-7 and at the dose of 300 IU from day 8 to the end of stimulation (maximal dose adjustment to 450 IU).
  Other interventions: conventional GnRH antagonist protocol and in vitro fertilization (IVF/ICSI) cycle
  Other Names: Elonva, Merional
  Arms: Corifollitropin alfa and menotropin
Drug: Follitropin alfa and lutropin alfa — Procedure: Ovarian stimulation is performed with daily 300 IU of Follitropin alfa and lutropin alfa starting on menstrual cycle day 2-3. Maximal allowed dose adjustment is 450 IU daily.
  Other interventions: conventional GnRH antagonist protocol and in vitro fertilization (IVF/ICSI) cycle.
  Other Names: Pergoveris
  Arms: Follitropin alfa and lutropin alfa

SUMMARY:
In an opened randomized study of women undergoing in vitro fertilization with expected suboptimal response to controlled ovarian stimulation (Poseidon Group 2b) investigators will examine clinical efficacy and safety of two stimulation protocols: Corifollitropin alfa (Elonva) in combination with menotropin (Merional) versus Follitropin alfa and lutropin alfa (Pergoveris).

DETAILED DESCRIPTION:
Patients, found eligible for the study, will be randomized (envelope method) into two arms in 1:1 ratio at the start of stimulation (menstrual cycle day 2-3, randomization day): Arm A - ovarian stimulation with Corifollitropin alfa in combination with menotropin; Arm B - ovarian stimulation with Follitropin alfa and lutropin alfa.

At the first day of controlled ovarian stimulation (COS) participants in the first group will receive a single injection of Corifollitropin alfa 150 mcg followed by daily menotropin administration at the dose of 150 international unit (IU) from stimulation day 1 to day 7 and at the dose of 300 IU from day 8 up to the end of stimulation.

Ovarian stimulation in group B will be performed with daily 300 IU of Follitropin alfa and lutropin alfa starting on menstrual cycle day 2-3.

For all subjects, a fixed dose of gonadotropin-releasing hormone (GnRH) antagonist will be injected daily as soon as one of the follicles reaches the ≥14 mm diameter and stopped one day before oocyte pick up (OPU); ovulatory dose of human chorionic gonadotropin (hCG) could be administered when at least one follicle reaches 16.5 mm in diameter.

Retrieved oocytes following fertilization (conventional IVF or ICSI) will be cultured to morula or blastocyst stage followed by ultrasound guided single or double embryo transfer (ET day, performed 4-5 days after OPU).

ELIGIBILITY:
Inclusion Criteria:

* Female age between 35-41 years;
* BMI 17,5-30 kg/m2;
* Expected suboptimal responders (according to Poseidon classification, 2016, Group 2b): patients with suboptimal ovarian reserve prestimulation parameters in terms of antimüllerian hormone (AMH) and antral follicle count (AFC): AFC 5-9, AMH ≥0.8 ng/mL;
* Early follicular phase follicle stimulating hormone (FSH) ≤15 IU/L;
* Presence of viable spermatozoa in partner's sperm;
* Signed informed consent.

Exclusion Criteria:

* Pre-existing medical condition preventing or interfering with IVF treatment: any clinically significant systemic disease; inherited or acquires thrombophilia and thromboembolism; endocrine or metabolic abnormalities; moderate or severe impairment of renal or hepatic function; any oncological diseases in anamnesis; known history of recurrent miscarriage, abnormal karyotype of both partners; currently active pelvic inflammatory disease;
* Abnormal IVF screening tests: Papanicolaou test, Syphilis, HIV 1&2, Hepatitis B, Hepatitis C, Chlamydia, and Gonorrhea;
* Presence of uterine pathology: Asherman's Syndrome, endometrial polyps, nodus form of adenomyosis or uterine fibroids ≥3 mm in diameter;
* Visualization of ovarian cysts ≥25 mm, endometriomas or hydrosalpinx;
* One or more follicles ≥8 mm on randomization day.

Ages: 35 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Number of cumulus-oocyte complexes (COCs) | 3-4 weeks after ET
  Number of COCs, obtained during oocyte pick up (OPU), after controlled ovarian stimulation (COS) in two protocols

SECONDARY OUTCOMES:
Duration of stimulation | 2-4 weeks after randomization
  total days of COS: from the first gonadotropins administration to ovulation triggering
Number of follicles at the end of stimulation | 2-4 weeks after randomization
  measured for follicles ≥17 mm and ≥14 mm
Dose adjustment frequency | 2-4 weeks after randomization
  number of participants with menopausal or recombinant human follicle stimulating hormone (FSH) dose increase
Number of participants with optimal or suboptimal response to COS | 2-4 weeks after randomization
  ≥ 5 COCs at at oocyte recovery day
Number of mature (MII) oocytes | 2-4 weeks after randomization
  assessment is done only for ICSI cycles at oocyte recovery day
Cycle cancellation rate | 6-7 weeks after randomization
  number of cancelled cycles during COS (no response), at OPU (premature ovulation, absence or degradation of COCs), during in vitro cultivation (fertilization failure, inadequate embryo quality) or due to other reasons (adverse events, ovarian hyperstimulation syndrome (OHSS), withdrawal)
Frequency of side reactions | 2-4 weeks after randomization
  number of patients with local reactions (redness, itching, swelling or pain) or abdominal discomfort evaluated using visual analogue scale at the end of COS and at ET day
Implantation rate | 3-4 weeks after ET
  ratio of the number of intrauterine gestational sacs to the number of transferred embryos
Clinical pregnancy rate | 5-6 weeks after randomization
  presence of intrauterine gestational sac at transvaginal ultrasound measured per embryo transfer

OTHER OUTCOMES:
Biochemical pregnancy rate | 3-4 weeks after ET
  positive ß-hCG test (≥30 IU/L) following ET without clinical pregnancy confirmation
Fertilization rate | 1 day after OPU
  number of two-pronuclear zygotes on day 1 after fertilization
Embryo quality | 3-5 days after oocyte recovery
  number of best and good quality embryos per transfer
Cost-effectiveness of COS | 6-7 weeks after randomization
  ratio of total cost of stimulation (on investigated drugs) to the number of patients with clinical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Alexdandr Gzgzyan, Prof, PhD, Principal Investigator — D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology
Locations (1):
- D.O. Ott Research Institute of Obstetrics, Gynecology, and Reproductology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ob'edkova KV, Kogan IY, Muller VC, Tapilskaya NI, Krikhely IO, Dzhemlikhanova LK, Abdulkadirova ZK, Mekina ID, Lesik EA, Komarova EA, Ishchuk MA, Gzgzian AM. IVF protocol efficacy in women with expected suboptimal response depending on ovary stimulation mode. Gynecol Endocrinol. 2021;37(sup1):44-48. doi: 10.1080/09513590.2021.2006526. PMID 34937512